CLINICAL TRIAL: NCT06726928
Title: SiREX-Stent for the Treatment of SymptOmatic Lateral VEnous Sinus Stenosis
Acronym: RESOLVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESOLVE
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Treatment of Symptomatic Lateral Sinus Stenosis; Treatment of Pulsatile Tinnitus Due tu Sinus Stenosis
Keywords: Pulsatile Tinnitus; Sinus vein stenosis
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Novel medical device
  Interventions: Device: Sinus Stenting

INTERVENTIONS:
Device: Sinus Stenting — Stenting of symptomatic sinus stenosis

SUMMARY:
The purpose of the study is to assess the efficacy, safety and the clinical benefit of the SiREX stent for the treatment of disabling pulsatile tinnitus due to stenosis of lateral sinus.

The study will enrol patients suffering from pulsatile tinnitus related to a lateral sinus stenosis lasting more than three months, and who want to be treated with lateral sinus stenting

DETAILED DESCRIPTION:
As there is currently no specifically developed and approved stent on the market for the treatment of symptomatic sinus stenosis, stenting has so far been performed with stents intended for carotid stenosis or peripheral treatment, which leads to considerable limitations. Because of stiff delivery systems (6F or bigger) progression inside the venous sinus is sometimes difficult. Furthermore, the length of such devices is often insufficient to cover the entire pathological segment and more than one device needs to be implanted in an overlaying manor (telescoping), which is accompanied with higher complication risks.

The objective of the study is to prove the efficacy and clinical safety of the new dedicated SiREX Stent with optimized technical features (smaller delivery system, longer lengths, reduced radial force), specially developed for the treatment of venous sinus stenosis. Pulsatile tinnitus is expected to disappear immediately after treatment with a stable effect during time.

ELIGIBILITY:
Inclusion Criteria:

* • Patient ≥ 18 years old

  * Disabling pulsatile tinnitus lasting for more than three months
  * Venous type: pulsatile tinnitus is interrupted by ipsilateral jugular vein compression
  * Lateral sinus stenosis visible on venous MRA or venous angio CT
  * Exclusion of other cause (excepted dehiscence of the lateral sinus related to the stenosis) of PT on MRI and on the temporal bone CT
  * Stenosis located on a dominant or codominant lateral sinus
  * Stenosis associated with a venous gradient of at least 3 mm Hg under general anesthesia (GA) in the absence of sinus dehiscence, or 2 mm Hg under GA if there is sinus dehiscence in a mastoid cell
  * Patients asking for the treatment of her/his pulsatile tinnitus
  * Patients accepting to receive the SiREX® Stent (instead of a carotid stent)
  * Written informed consent

Exclusion Criteria:

* Non-pulsatile tinnitus or pulsatile tinnitus unrelated to lateral sinus stenosis
* Stenosis with gradient < 2 mm Hg in the absence of associated lateral sinus dehiscence
* Any contraindication for treatment according to Instructions for Use:

  * Patients in whom the size of the venous vessel section to be treated does not lie within the range indicated for the stent.
  * Patients for whom angiography shows that the anatomic morphology is not suitable for endovascular treatment due to severe vessel tortuosity or stenosis.Patients who were not pre-treated with antiplatelet agents prior to the procedure.
  * Patients in whom treatment with antiplatelet agents and/or anticoagulants is contraindicated.
  * Patients with an acute subarachnoid haemorrhage.
  * Patients with an active bacterial infection.
  * Patients who are hypersensitive to nickel-titanium.
* Pregnant or breastfeeding woman
* Subject is participating in another clinical study
* Patients with a life-threatening event in the last 6 months
* Patients with a life expectancy under 12 months
* Known, severe comorbidities, which will likely influence carrying out of the follow-up visits (cancer, alcohol/drug abuse or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Disappearance of pulsatile tinnitus at 90 (± 20) days | 90 days
  Disappearance of pulsatile tinnitus at 90 (± 20) days after resolving of the lateral sinus stenosis with SiREX Stent

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lariboisière, Paris, France